CLINICAL TRIAL: NCT03967093
Title: A Phase 1 Safety Study of BXQ-350 Administered as a Single Agent by Intravenous Infusion in Children and Young Adults With Relapsed Solid Tumors, Including Recurrent Malignant Brain Tumors
Brief Title: A Study of BXQ-350 in Children and Young Adults With Relapsed Solid Tumors
Acronym: KOURAGE
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Bexion will not move forward with the Part 2 expansion portion of the trial in order to focus resources on the further development of BXQ-350 as an earlier treatment measure in the pediatric population.
Sponsor: Bexion Pharmaceuticals, Inc. (Industry)
Collaborators: CTI Clinical Trial and Consulting Services (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BXQ-350.AB
Record Dates: First submitted 2019-05-21; First posted 2019-05-30 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Neoplasms
Keywords: solid tumor; brain tumor; DIPG; ependymoma
MeSH Terms: conditions — Neoplasms; Brain Neoplasms; Ependymoma

STUDY DESIGN:
Intervention Model Description: Part 1 dose escalation - sequential cohorts of patients will be treated with escalating doses of BXQ-350 until the maximum tolerated dose (MTD) is established, or in the absence of a maximum administered dose, the highest planned dose level.
  Part 2 - patients will be enrolled and administered BXQ-350 at the Part 1 MTD or at the highest planned dose level
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1 Dose Escalation: Safety and Tolerance (Experimental): Sequential cohorts of patients with relapsed solid tumors, including malignant brain tumors, will be treated with escalating doses of BXQ-350 until the maximum tolerated dose (MTD) is established, or in the absence of a maximum administered dose (MAD), the highest planned dose level (3.2 mg/kg) is reached.
  Interventions: Drug: BXQ-350
- Part 2: Ependymoma Patients (Experimental): Cohort of patients with recurrent ependymoma will be enrolled and administered BXQ-350 at the MTD determined in Part 1 or at 3.2 mg/kg if the MAD is not reached.
  Interventions: Drug: BXQ-350
- Part 2: Brain Tumor Patients (Experimental): Cohort of patients with recurrent malignant brain tumors will be enrolled and administered BXQ-350 at the MTD determined in Part 1 or at 3.2 mg/kg if the MAD is not reached.
  Interventions: Drug: BXQ-350
- Part 2: DIPG Patients (Experimental): Cohort of patients with recurrent diffuse intrinsic pontine glioma (DIPG) will be enrolled and administered BXQ-350 at the MTD determined in Part 1 or at 3.2 mg/kg if the MAD is not reached.
  Interventions: Drug: BXQ-350
- Part 2: Other Solid Tumor Patients (Experimental): Cohort of patients with relapsed non-central nervous system (CNS) solid tumors will be enrolled and administered BXQ-350 at the MTD determined in Part 1 or at 3.2 mg/kg if the MAD is not reached.
  Interventions: Drug: BXQ-350

INTERVENTIONS:
Drug: BXQ-350 — BXQ-350 is a novel anti-neoplastic therapeutic agent configured from two components: Saposin C (SapC), an expressed (human) lysosomal protein, and the phospholipid dioleoylphosphatidyl-serine (DOPS), a phospholipid located on cell membranes (clinical formulation BXQ-350). BXQ-350 is administered by intravenous (IV) infusion over a minimum of six 28-day cycles.
  Other Names: SapC-DOPS

SUMMARY:
This study will evaluate the safety of BXQ-350 and determine the maximum tolerated dose (MTD) in children and young adults with relapsed solid tumors, including recurrent malignant brain tumors. All patients will receive BXQ-350 by intravenous (IV) infusion. The study is divided into two parts: Part 1 will enroll patients at increasing dose levels of BXQ-350 in order to determine the MTD. Part 2 will use the MTD to further assess the safety of BXQ-350 as well as preliminary anti-tumor activity.

DETAILED DESCRIPTION:
BXQ-350 is a novel anti-neoplastic therapeutic agent configured from two components: Saposin C (SapC), an expressed (human) lysosomal protein, and the phospholipid dioleoylphosphatidyl-serine (DOPS), a phospholipid located on cell membranes (clinical formulation BXQ-350). Given via intravenous (IV) infusion, data indicate that the agent exhibits the propensity to enter the body and brain, target cells in the tumor mass, and induce cell death.

The study is divided into 2 parts:

Part 1: Dose Escalation and Safety - Sequential cohorts of patients 1-30 years of age with relapsed solid tumors, including recurrent malignant brain tumors will be treated with escalating doses of BXQ-350 until the MTD is established, or in the absence of a Maximum Administered Dose, the highest planned dose level is reached.

Part 2: Safety and Preliminary Anti-tumor Activity - Patients will be enrolled into one of four cohorts and administered BXQ-350 at the established MTD or at the highest planned dose level. The four cohorts will consist of: recurrent ependymoma, recurrent malignant brain tumor, recurrent Diffuse Intrinsic Pontine Glioma (DIPG), and relapsed non-central nervous system (non-CNS) solid tumor.

ELIGIBILITY:
Inclusion Criteria:

* Each subject must meet the following criteria:

  1. Provide signed, written informed consent prior to the initiation of any study-specific procedures (Consent from Guardians for minor children and patient assent according to Institution and Institutional Review Board (IRB) standards)
  2. Are male or female aged ≥ 1 to 30 years
  3. Have histologically or cytologically confirmed relapsed solid tumor cancer, including recurrent malignant brain tumors, for which there is no further standard therapy or when standard therapy is contraindicated • Recurrent malignant brain tumors: must have shown unequivocal evidence for recurrence or progression by MRI scan or must have histologically proven tumor recurrence • Recurrent malignant brain tumors: must have previously received standard of care treatment at initial diagnosis (radiation and/or chemotherapy)

     * Recurrent malignant brain tumors receiving glucocorticoid therapy: must be on stable or decreasing equivalent daily dose of glucocorticoids for 2 weeks (14 days) prior to dose assignment
     * Recurrent embryonal tumors or atypical teratoid rhabdoid tumors (AT/RT): must have previously received standard of care therapy including either chemotherapy and radiation therapy or high dose chemotherapy with autologous hematopoietic stem cell support
     * Grade II or III recurrent ependymoma, including RELA fusion-positive ependymoma: must have previously received radiation therapy
  4. Have measurable or non-measurable disease per RECIST v1.1 for relapsed solid tumors, RRC for recurrent malignant brain tumors, and INRC for recurrent neuroblastomas
  5. Have Lansky (age 1 - 15) / Karnofsky (age ≥ 16) Performance Score of >50 or Eastern Cooperative Oncology Group Performance Status (ECOG PS) (age ≥ 18) of 0 - 2
  6. Have acceptable liver function defined as:

     * Total serum bilirubin ≤ 1.5 × upper limit of normal (ULN) for the study site (in subjects with known Gilbert Syndrome, total bilirubin ≤ 3 × ULN, with direct bilirubin ≤ 1.5 × ULN)
     * Aspartate Transaminase (AST), Serum Glutamic Oxaloacetic Transaminase (SGOT), Alanine Transaminase (ALT), Serum Glutamic-Pyruvic Transamine (SGPT) ≤ 3 × ULN (if liver metastases are present, then ≤ 5 × ULN is allowed)
     * Serum albumin ≥ 3 g/dL
  7. Have acceptable renal function defined as:

     * Creatinine clearance or radioisotope glomerular filtration rate (GFR) ≥70 mL/min/1.73m² or a maximum serum creatinine (mg/dL)* based on age/gender as follows:

       1 to < 2 years: 0.6 (male); 0.6 (female)

       2 to < 6 years: 0.8 (male); 0.8 (female)

       6 to < 10 years: 1 (male); 1 (female)

       10 to < 13 years: 1.2 (male); 1.2 (female)

       13 to < 16 years: 1.5 (male); 1.4 (female)

       ≥ 16 years: 1.7 (male); 1.4 (female)

       * Threshold creatinine values derived from the Schwartz formula for estimating GFR utilizing child length and stature data published by the CDC (Schwartz 2009)
  8. Have acceptable bone marrow function defined as:

     * Absolute neutrophil count (ANC) ≥ 750 cells/mm3
     * Platelet count ≥ 75,000 cells/mm3
     * Hemoglobin > 9.0 g/dL
  9. Have acceptable coagulation parameters defined as:

     * International normalized ratio (INR) ≤ 2 × ULN
     * Activated partial thromboplastin time (aPTT) within normal limits
     * Chronic/prophylactic anticoagulation for a distant thrombus that occurred ≥3 months ago is allowed
  10. Have a negative serum pregnancy test result at screening (for females of child bearing potential (FCBP); not applicable to subjects who are unable to become pregnant, including those with tubal ligation, bilateral oophorectomy and/or hysterectomy)
  11. FCBP and male subjects whose sexual partner(s) are FCBP must agree to abstain from heterosexual activity or use a double barrier method of contraception (e.g., condom and occlusive cap with spermicide) or highly effective contraception (intrauterine device or system, established hormonal contraceptive methods on a stable dose from the time of the last menstrual cycle, or vasectomized partner with confirmed azoospermia) from the time of study entry to 1 month after the last day of treatment

Exclusion Criteria:

- Subjects must not meet any of the following criteria:

1. Have a concurrent or second malignancy
2. Have lymphoma
3. Have Grade I ependymoma
4. Relapsed solid tumors: have symptomatic brain metastases or leptomeningeal disease
5. Relapsed solid tumors: have received

   * anticancer therapies within 2 weeks prior to dose assignment (including radiation therapy, cytotoxic agents, targeted agents or endocrine therapy)
   * myelosuppressive agents within 3 weeks prior to dose assignment
   * monoclonal antibodies within 4 weeks prior to dose assignment
   * growth factors within 2 weeks of dose assignment
   * other immunotherapy (tumor vaccine, cytokines) within 4 weeks of dose assignment
6. Recurrent malignant brain tumors: have received

   * anticancer therapies including: radiation therapy to current site of disease within 3 weeks dose assignment; targeted agent therapy within 2 weeks of dose assignment; nitrosoureas within 6 weeks of dose assignment; procarbazine within 3 weeks of dose assignment; other cytotoxic agents withing 4 weeks of dose assignment
   * myelosuppressive agents within 4 weeks prior to dose assignment
   * monoclonal antibodies within 4 weeks prior to dose assignment
   * other immunotherapy (tumor vaccine, cytokines, or growth factor) within 2 weeks prior to dose assignment
7. Have not recovered from toxicity of prior therapy defined as a return to ≤ grade 1 at the time of dose assignment, graded according to CTCAE v5.0 (excluding alopecia, neuropathy, and lymphopenia)
8. Have had major surgery other than a minor outpatient procedure within 28 days prior to dose assignment or have not recovered from major side effects of the surgery if more than 4 weeks have elapsed since surgery
9. Have poorly controlled hypertension despite the use of antihypertensive agents defined as blood pressure ≥95th percentile for age and weight or >160/90 on at least 2 repeated determinations on separate days within 2 weeks (14 days) prior to initiation of screening
10. Have a history of cardiac dysfunction including any of the following:

    * Myocardial infarction within 6 months prior to initiation of screening
    * History of documented congestive heart failure (New York Heart Association functional classification III-IV, see Appendix 6) within 6 months prior to initiation of screening
    * Active cardiomyopathy
    * Electrocardiogram (ECG) with QTc >480 msec at screening
    * Echocardiogram with ejection fraction <50% or a decrease in the left ventricular shortening fraction to <27%
11. Have a known history of Human Immunodeficiency Virus (HIV) seropositivity
12. Have active (acute or chronic) or uncontrolled severe infections
13. Have active poor wound healing (delayed healing, wound infection or fistula)
14. Have evidence of active clinically significant bleed (e.g., gastrointestinal bleed, hemoptysis, or gross hematuria) at initiation of screening
15. Are pregnant or nursing (lactating), where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive serum human chorionic gonadotropin (hCG) laboratory test
16. Have received prior treatment with any investigational drug within 28 days prior to dose assignment
17. Have other concurrent severe and/or uncontrolled medical condition that would, in the site Investigator's judgment contraindicate the subject's participation in the clinical study

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-01-03 (Actual); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events as Assessed by CTCAE v5.0 | 6 months
  To determine the safety of BXQ-350 in children and young adults with relapsed solid tumors, including recurrent malignant brain tumors, as evidenced by the incidence of treatment emergent adverse events assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Part 1 - Maximum Tolerated Dose | 6 months
  To determine the maximum tolerated dose (MTD) of BXQ-350, when given as a single agent at escalating doses, according to the investigational product (IP) related dose limiting toxicities (DLTs) in children and young adults with relapsed solid tumors, including recurrent malignant brain tumors
Part 2 - RECIST | 6 months
  To assess the preliminary antitumor activity of BXQ-350, given as a single agent at the MTD, or highest planned dose level (DL), 3.2 mg/kg, in the absence of a Maximum Administered Dose (MAD). Antitumor activity is defined as maximal radiological response during treatment using:
  • Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (v1.1) criteria for relapsed solid tumors
Part 2 - RANO | 6 months
  To assess the preliminary antitumor activity of BXQ-350, given as a single agent at the MTD, or highest planned dose level (DL), 3.2 mg/kg, in the absence of a Maximum Administered Dose (MAD). Antitumor activity is defined as maximal radiological response during treatment using:
  • Radiographic Response Criteria (RRC) for recurrent malignant brain tumors
Part 2 - INRC | 6 months
  To assess the preliminary antitumor activity of BXQ-350, given as a single agent at the MTD, or highest planned dose level (DL), 3.2 mg/kg, in the absence of a Maximum Administered Dose (MAD). Antitumor activity is defined as maximal radiological response during treatment using:
  • International Neuroblastoma Response Criteria (INRC) for recurrent neuroblastomas

SECONDARY OUTCOMES:
Progression-Free Survival (PFS-6) | 6 months
  · To evaluate progression-free survival at 6 months (PFS-6) in subjects with relapsed solid tumors, including recurrent malignant brain tumors
Time to Response | 6 months
  · To evaluate time to response, and duration of response in subjects with relapsed solid tumors, including recurrent malignant brain tumors
Duration of Response | 6 months
  · To evaluate duration of response in subjects with relapsed solid tumors, including recurrent malignant brain tumors

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No